CLINICAL TRIAL: NCT01492478
Title: Psychobiological Characterization of Depression in Hepatitis C
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centro Hospitalar Lisboa Norte (Other)
Responsible Party: Principal Investigator, David Pires Barreira, Dr., Centro Hospitalar Lisboa Norte
Other Study IDs: 39772
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Depression; Hepatitis c
MeSH Terms: conditions — Depression; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to do an evaluation of the clinical profile of depression in HCV patients (newly diagnosed and treatment naïve), and in these same individuals, 24 weeks after the beginning of IFN+Ribavirin therapeutics (n=100). To characterize depression associated to HCV with and without interferon (IFN), the investigators will use clinical, behavioral, biochemical and genetic markers, and to distinguish their different symptomatologic dimensions.

The control group will be composed by 100 individuals with Major Depression diagnosis, and not from the general population, because the investigators are not trying to study the incidence of depression in general population, but to characterize the clinical profile of patients with HCV (IFN+Ribavirin) compared to major depression.

Thus, the investigators will total 300 evaluations in 200 individuals, 100 from each group, and considering that the clinical group will be evaluated before the therapeutics and re-evaluated 24 weeks after its beginning.

Hypotheses

1. Depression in individuals affected by HCV is associated to genetic vulnerability.
2. Genetic vulnerability increases the risk of depression when IFN therapeutics is used.
3. Depression associated to infection by HCV presents a symptomatological profile that is different from general depression, which is maintained with IFN therapeutics.
4. A higher state of depression in the beginning of a treatment, if not treated, is a risk factor to abandoning therapeutics.
5. When comparing genders, women present a more severe symptomatological profile than men.

DETAILED DESCRIPTION:
The World Health Organization (WHO) estimates that about 3% of the world population (170 million people) is infected with the hepatitis C virus (HCV). In Portugal, there were an estimated 150.000 cases, of which only 10% have confirmed diagnosis. The disease's potential of evolution towards chronicity, hepatic cirrhosis and hepatocellular carcinoma, makes this the main indicator for liver transplant. Besides the natural history of this disease and the burden that it causes in the economy, these individuals frequently present neuropsychiatric symptoms like fatigue, anxiety, depression and cognitive disorders.

Among these, depression stands out for its enormous impact on individuals and society. Reaching higher than 15%, this will be the second most prevailing disease in the world by 2020, according to WHO predictions.

Regarding neuropsychiatric symptoms, one can identify two distinctive patterns in its relation with HCV infection. On one hand, individuals with chronic hepatitis C have higher prevalence of psychiatric disorders, including depression. On the other hand, individuals with psychiatric records present higher HCV infection rates than the average population.

A combined therapeutics of pegylated interferon (IFN) and ribavirin is used in these patients as the standard treatment, and proves to be a fundamental and consensual intervention for a favorable change in the natural history of the disease. However, this treatment is associated with a high number of adverse reactions like: "influenza-like" symptoms, irritability, insomnia, fatigue and loss of appetite. Apart from these, neuropsychiatric symptoms (specially depression, and sometimes with suicidal ideation), are among the most common secondary effects in therapeutics with IFN, being one of the main causes why patients interrupt their treatment. It is noteworthy that, up to a certain extent, psychopathologic symptoms (depression, cognitive disorders) may be associated to HCV infection, even without an interferon treatment, and may be related to direct HCV neurotoxicity.

This symptomatology negatively affects the individual's perceived quality of life, its general functioning, work capacities, overall well-being and quality of life. Furthermore, therapeutic used in HCV treatment is associated to impairment in all of these dimensions.

Over the last years, there has been an increase in the research of the mechanisms that are likely to be responsible for the most serious collateral effects associated to this therapeutics, specially in cognitive disorders and depression cases.

IFN induces changes in the endocrine function (hypothalamic-pituitary-adrenal axis) and in neurotransmission activity (specially serotonin and dopamine).

The mechanism by which depression is induced by IFN is still being researched and it is, very likely, multifactorial. Several studies suggest that an imbalance between Th1 and Th2 cytokine or pro-inflammatory and anti-inflammatory cytokine may have an important role in the modulation of cellular responses in the brain during psychological stress and psychological disorders. A recent study, and in agreement with the growing literature about the relation between inflammatory cytokine and the serotonin pathways (5-HT), shows that IFN can affect the expression of serotonergic 1A receptors (5-HT1A), which is consistent with what is observed in depressed individuals. IFN also reduces the levels of peripheric tryptophan, an effect that is correlated to depression.

Several studies and meta-analysis have implied polymorphisms in the promotor region of the serotonin transporter gene (5-HTT), so called 5-HTTLPR, in response to treatment with selective serotonin reuptake inhibitors in patients with major depression. In the same way, 5-HTTLPR seems to be associated with a higher occurrence of this disease during IFN treatment. This alludes to an association between exposition to inflammatory cytokine (IFN) and the existence of some variability in the 5-HTTLPR of major depression.

The cytokine therapy model has been used to study physiopathology of depression induced by cytokine. Here, it is worth distinguishing two behavioral syndromes with different phenomenology and response capacity to antidepressants in patients that became depressed with cytokine. On one hand, mood and cognitive syndrome, characterized by typical depression symptoms, like depressed mood, anxiety, irritability, memory and attention disorders, which usually develops between the first and the third month of IFN treatment in vulnerable patients. On the other hand, a neurovegetative syndrome, manifested by symptoms of fatigue, psychomotor slowness, anorexia and changes in sleep patterns, develops relatively early (after two weeks of treatment with IFN) and, in a large number of individuals remains until later stages of the treatment.

In terms of the response capacity to antidepressants, mood and cognitive syndrome have had a very good effectiveness when pre-treated with paroxetine (an selective serotonin reuptake inhibitor), whereas neurovegetative syndrome has not had any response to it. Thus, this data suggests that different physiopathological pathways may be connected to the development of specific symptomatic dimensions, including mood/cognitive symptoms versus neurovegetative symptoms, in the context of the cytokine activation system.

However, the available literature about HCV associated depression is wide and contradictive. For instance, the percentages of depression incidence in this population vary between 15% and 60%, depending on how many samples and methodologies are used. This way, it seems pertinent to perform a research project that focuses characterization of the depressive profile, not only from the clinical point of view, but also using biochemical and genetics markers in this population.

Thus, it is the intention of this work to pursue a better understanding of the neuropsychiatric symptoms associated to hepatitis C, depression in particular. This way we intend to achieve relevant contributes, on a preventive and therapeutic approaches to this population.

ELIGIBILITY:
Inclusion Criteria:

* minimum education;
* ages between 18 and 65 years old;
* with diagnosis of Hepatitis C for at least 6 months, newly diagnosed and treatment naive;
* and diagnosis of Major Depression for the control group.

Exclusion Criteria:

* consumption of opiates, cocaine or other recreational drugs in the 6 months prior to the beginning of the research;
* use of anti-inflammatory drugs and antidepressants;
* history of neurological, infectious or tumoral pathology, at SNC level;
* severe physical deterioration incompatible with the situation being evaluated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are selected in the context of hospital consultancies (Viral Hepatitis Consultancies at the Hospital de Santa Maria; Psychiatric Consultancies at the Hospital de Santa Maria) after informing, requesting voluntary cooperation, confidenciality assurance and with request of informed consent signature, submitted and approved by the hospital's ethics committee
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Pires Barreira, Dr., Principal Investigator — Centro Hospitalar Lisboa Norte
Locations (1):
- Faculty of Medicice of Lisbon, Lisbon, Portugal